CLINICAL TRIAL: NCT06163573
Title: Treatment of Patellofemoral Osteoarthritis With Nasal Chondrocyte-based Engineered Cartilage Implantation in a Randomized, Controlled, Multi-center Phase II Clinical Trial
Brief Title: Treatment of Patellofemoral Osteoarthritis With Engineered Cartilage.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other); Clinical Trial Unit, University Hospital Basel, Switzerland (Other); University Hospital Wurzburg (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-508640-21-00
Record Dates: First submitted 2023-11-20; First posted 2023-12-11 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Patellofemoral Osteoarthritis
Keywords: Nasal chondrocytes; Tissue engineering; Knee cartilage; Patellofemoral osteoarthritis

STUDY DESIGN:
Intervention Model Description: Experimental group: biological: Autologous nasal chondrocytes and ECM proteins Control group: Platelet rich plasma injections
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-TEC (Experimental): N-TEC is based on autologous nasal chondrocytes expanded and further cultured on type I/III collagen membranes for 2 weeks to allow cells to produce extracellular matrix containing cartilage specific proteins. The IMP is implanted in the knee at the patellofemoral joint.
  Interventions: Biological: N-TEC
- Platelet Rich Plasma (Active Comparator): Total of 3 injections of about 5 ml each of platelet rich plasma (PRP), autologous Conditioned Plasma ACP®, Arthrex, one injection per week for three consecutive weeks.
  Interventions: Biological: Platelet rich plasma

INTERVENTIONS:
Biological: N-TEC — Implantation of an autologous tissue engineered cartilage graft in the patellofemoral joint for treatment of osteoarthritis.
  Other Names: Engineered cartilage graft
  Arms: N-TEC
Biological: Platelet rich plasma — Injection of an autologous Conditioned Plasma ACP® on the basis of one injection per week for three consecutive weeks.
  Conditioned Plasma ACP®, Arthrex, one injection per week for three consecutive weeks.
  Other Names: PRP
  Arms: Platelet Rich Plasma

SUMMARY:
The purpose of this investigator-initiated study is to assess the efficacy of treating patellofemoral osteoarthritis with an Advanced Therapy Medicinal Product (ATMP), autologous nasal chondrocyte tissue engineered cartilage (N-TEC), in comparison with a standard therapy using platelet rich plasma injections.

The engineered cartilage graft is obtained by culturing expanded autologous nasal chondrocytes within a collagen type I/III membrane.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is one of the most common causes for pain and disability with over 260 million people affected worldwide. Recent studies found that knee OA often starts in the patello-femoral compartment of the knee (PFOA) and is diagnosed in ~39% of people with knee pain aged above 30 years. Thus, PFOA and progression to full OA plays a crucial role in the reduction of quality of life of many people and in the raise of healthcare costs.

The goal of this phase II trial is to (i) evaluate the efficacy of autologous Nasal Chondrocytes Tissue Engineered Cartilage (N-TEC) in comparison to an active comparator (Platelet Rich Plasma (PRP) injections) based on patients' self-assessed outcome scores (Knee Osteoarthritis Outcome Score (KOOS Pain), and to (ii) verify tissue regeneration as the postulated mode of action and thus the disease-modifying properties of the graft, as previously indicated in animal studies (x-ray, MRI). This proposed phase II trial will evaluate whether N-TEC improves the clinical efficacy, leading to an increase of at least 15 points higher in the main primary outcome (KOOS (pain) change at 24 months) than the comparator group. Secondary endpoints will include amongst others KOOS subscales (symptoms, pain, activity of daily living (ADL), sports, Quality of Life (QOL)), Kujala Anterior Knee Pain Scale, Western Ontario and McMaster Universities Osteoarthritis score (WOMAC), Marx Activity Rating Scale (MARS) and EQ-5d assessment at 6, 12 and 24 months compared to baseline and between groups. Further secondary endpoints will be the number of subjects non-responding to treatment (i.e., improvement in KOOS Pain below 13 units on a scale of 0-100) and treatment failures (deterioration of more than 13 points compared to baseline or switching to other regenerative treatments or joint replacement to evaluate efficacy). Adverse events will be recorded during the full course of the trial to assess safety. This will require enrolling a total of 75 patients in a multicenter, prospective study involving 9 clinical centers.

ELIGIBILITY:
Inclusion Criteria:

* Patient age is ≥18 and ≤ 65 years at time of screening.
* Symptomatic PFOA grade 1-3 according to Iwano Classification
* Chondropathy Grade 3-4 according to ICRS classification of the patella, trochlea femoris or both
* Baseline score of <60 on the KOOS Pain subjective knee evaluation.
* Free range of motion of the affected knee joint or ≤ 5° of extension loss and minimum 125° flexion.
* Patient is willing and able to give written informed consent to participate in the study and to comply with all study requirements, including attending all follow-up visits and assessments and to complete postoperative rehabilitation regimen.
* Minimum values for women: Haemoglobin 120g/l, Platelets 150G/l, INR<1.3
* Minimum values for men: Haemoglobin 140g/l, Platelets 150G/l, INR<1.3
* Non-surgical standard of care options except for PRP have been exhausted.

Exclusion Criteria:

* Patient is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol or in a dependency or employment with the sponsor.
* Patient is unable to understand the patient information
* Patient is unable to undergo magnetic resonance imaging (MRI)
* Prior surgical treatment of the target knee within 12 months (Note: prior diagnostic arthroscopy with debridement and lavage are acceptable within 12 months).
* Radiologically apparent degenerative joint disease of the tibiofemoral joint as determined by X-ray (Kellgren and Lawrence grade > 2) or MRI or pain in the tibiofemoral joint as assessed by clinical examination
* Patient has excessive varus or valgus deformity (>5°)
* Patient had a patellar dislocation in the afflicted knee in the last 2 years.
* Patient has a symptomatic meniscus lesion (or removal exceeding ½), as indicated by clinical examination (joint line tenderness and McMurray test positive) and MRI.
* Patient has a body mass index (BMI) >35 kg/m2.
* Patient has chronic rheumatoid arthritis, and/or infectious arthritis
* Any concomitant painful or disabling disease of the spine, hips, or lower limbs that would interfere with evaluation of the afflicted knee.
* Patient has a known immunological suppressive disorder or is taking immunosuppressives.
* Patient had any intra-articular injections into the affected knee within the last 3 months before baseline visit
* Instability of anterior, posterior collateral ligaments
* The patient has a HIV/AIDS infection. (regulatory requirement)
* The patient has an acute Treponema pallidum (syphilis) infection. (regulatory requirement)
* The patient has an active hepatitis B or C infection with verified antigens. Patients with a cured hepatitis B or C infection and/or verified antibodies are not excluded. (regulatory requirement)
* Patient is pregnant, breast feeding or anticipates becoming pregnant within 24 months after surgery.
* Patient is currently participating or has participated in any other clinical study within 3 months prior to the screening visit.
* Patient has known current or recent history of illicit drug or alcohol abuse or dependence defined as the continued use of alcohol or drugs despite the development of social, legal or health problems.
* Patient has any other condition, which, in the opinion of the investigator, would make the patient unsuitable for the study.
* Any known allergies, especially for porcine collagen, penicillin or streptomycin (manufacturing)
* patients with increased anesthesiological and surgical risks (e.g. known or predicted difficult airway, myocardial infarction <60 days prior to surgery)
* patients with increased bleeding risk (e.g. coagulopathies)
* patients on anticoagulants whose anticoagulant therapy cannot be interrupted as appropriate to the given agent(s) and underlying condition
* Patients with any active infections

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) for pain | 24 months
  mean change in Knee Injury and Osteoarthritis Outcome Score for pain from baseline to 24 months between groups Minimum score: 0 Maximum score :100 (higher score means no knee problems)

SECONDARY OUTCOMES:
Biovigilance | until 24 months
  Number of adverse events, adverse reactions based on severity, expectedness and relationship to treatment.
Knee Injury and Osteoarthritis Outcome questionnaire | until 24 months
  patient self reported questionnaire for symptoms, activity of daily life, sports and quality of life Minimum score: 0 Maximum score: 100 (higher score means no knee problems)
Iwano classification | until 24 months
  Osteoarthritis grade determined based on X-rays according to Iwano classification (grades 1 to 4).
Kellgren Lawrence classification | until 24 months
  Osteoarthritis grade determined based on X-rays according to Kellgren Lawrence classification (grades 1 to 4).
MOCART score | until 24 months
  Magnetic Resonance Imaging (MRI) of Cartilage Repair Tissue (MOCART) score: radiological evaluation of repair tissue. Minimum score:0; maximum score: 100.
Kujala self reported questionnaire | until 24 months
  Anterior Knee Pain scale. Minimum score: 0 Maximum score: 100 (no knee problems)
EQ5d questionnaire | until 24 months
  patient self reported questionnaire including five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
  Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score | until 24 months
  Self reported questionnaire to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints.
  The instrument contains 24 items measuring 3 sub-scales: physical function (17 items), pain (5 items), and stiffness (2 items).
Visual Analogue Scale | Unitl 24 months
  The VAS is used by patients to assess pain based on a numbered scale going from 0 (no pain) to 10 (maximal pain).
Global Rating Of Change (GROC) likert scale | until 24 months
  Widely used score to assess whether the patient condition has gotten worse, better, or stayed the same and to quantify the magnitude of that change. Minimum score: -5 ; maximal score: +5.
Marx Activity Rating Scale (MARS) score | until 24 months
  This activity-related patient-reported outcome measure is widely used to assess the activity of a patient after treatment of the knee. It assesses how often the patient performs activities (running, cutting, deceleration and pivoting) in his healthiest and more active state. Minimum score: 0; maximum score: 16
Number of non responders | Until 24 months
  Number of treated patients showing an improvement in KOOS Pain below 13 on a scale of 0 to 100 after 24 months compared to baseline.
Number of treatment failures | Until 24 months
  Treatment failures are treated patients who had to switch to an alternative surgical regenerative treatment or knee replacement. This clinical deterioration is defined as reduction in the KOOS score of > 13 after 24 months compared to baseline.
MRI Osteoarthritis Knee Score (MOAKS) | Until 24 months
  MRI Osteoarthritis Knee Score (MOAKS) is a semi quantitative score used to assess the severity and progression of osteoarthritis in the knee using magnetic resonance imaging (MRI). It evaluates various features like osteophytes, bone marrow lesions, and cartilage loss, providing a detailed picture of the disease's status.

OTHER OUTCOMES:
Activity level | Until 24 months
  Patients will wear activity trackers for defined time periods to determine their activity level and assess if there is a correlation between the activity level and the clinical outcome.
Quality-adjusted life-years (QALY) outcome | Until 24 months
  Quality-adjusted life-years (QALY) is a measure of health outcome that combines the quantity and quality of life into a single value. It represents the value of an individual's health. QALY is used in cost-effectiveness analyses to compare the value of different healthcare interventions.
One Leg Hop test | Until 24 months
  The One Leg Hop test will be performed after patients had followed the physiotherapy program. This functional movement assessment is used to evaluate lower limb strength, power, and neuromuscular control. It involves hopping on one leg as far as possible and landing on the same leg while maintaining balance.
Y Balance test | Until 24 months
  The Y-Balance Test will be performed after patients had followed the physiotherapy program. It is a standardized test for assessing dynamic balance and movement quality, particularly in the lower extremities. It is used to assess injury risk and support post-injury rehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Mumme, Dr, Principal Investigator — University Hospital, Basel, Switzerland
Locations (9):
- Poliklinika Ivković, Zagreb, Croatia
- Germany (2):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Orthopädische Klinik König-Ludwig-Haus, Würzburg
- Switzerland (6):
  - University Hospital Basel, Basel
  - Crossklinik, Basel
  - Inselspital, Bern
  - Hôpitaux universitaires de Genève, Geneva
  - Ospedale Regionale di Lugano, Lugano
  - Sportclinic, Klinik Hirslanden, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seitz S, Lehoczky G, Wixmerten A, Schuster-Amft C, Miot S, Shrestha K, Schaedelin S, Martin I, Mumme M. Treatment of patellofemoral osteoarthritis with nasal chondrocyte-based engineered cartilage implantation in a randomised, controlled, multicentre phase II clinical trial: protocol for a randomised controlled trial. BMJ Open. 2025 Aug 21;15(8):e106140. doi: 10.1136/bmjopen-2025-106140. PMID 40840982